CLINICAL TRIAL: NCT03530475
Title: Diagnostic Accuracy of Doppler Ultrasound and Role of Uterine Artery Doppler in Cases of Placenta Accreta
Brief Title: Diagnostic Accuracy of Doppler Ultrasound and Role of Uterine Artery Doppler
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, hala nabil, principle investigator, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 5000
Record Dates: First submitted 2018-05-07; First posted 2018-05-21 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Placenta Accreta
MeSH Terms: conditions — Placenta Accreta | interventions — Ultrasonography, Doppler

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placenta previa (Active Comparator): cases diagnosed as placenta previa diagnosed by ultrasound and doppler
  Interventions: Diagnostic Test: ultrasound and doppler
- placenta accreta (Active Comparator): placenta previa diagnosed as placenta accreta by ultrasound and doppler
  Interventions: Diagnostic Test: ultrasound and doppler

INTERVENTIONS:
Diagnostic Test: ultrasound and doppler — • Ultrasound examination (2D gray scale and color doppler )
  1. Confirming the presence of placenta previa 2,To assess the possibility of concomitant placenta accreta (Sonographic findings that have been associated with placenta accreta (1) Loss of normal hypoechoic retroplacental zone (2) Multiple vascular lacunae (irregular vascular spaces) within placenta, (3) Blood vessels or placental tissue bridging uterine-placental margin, myometrial-bladder interface, or crossing uterine serosa1 (4) Retroplacental myometrial thickness of 1 mm (5) Bladder wall interruption (6) Presence of placental bulge (7) Utero-vesical hypervascularity (8) presence of lacunae feeder vessels.
  3. Assessment of uterine artery Doppler in different cases of placenta previa.
  . Documentation of the operative findings during cesarean section and/or cesarean hysterectomy procedures.
  Histopathological examination of the hysterectomy specimens to assess the degree of myometrial invasion.

SUMMARY:
This study will be conducted on (100) pregnant women diagnosed as placenta previa by ultrasonography and are candidates for either emergency or elective repeated cesarean section or hysterectomy (if the diagnosis of placenta accreta is confirmed).

All of those patients are presenting during the period of may 2018 to july 2018 to Kasr-Al Ainy Obstetrics outpatient clinic or casualty department during their 3rd trimester.

All of them will be assorted according to certain inclusion and exclusion criterions as follow:

DETAILED DESCRIPTION:
This study will be conducted on (100) pregnant women diagnosed as placenta previa by ultrasonography and are candidates for either emergency or elective repeated cesarean section or hysterectomy (if the diagnosis of placenta accreta is confirmed).

Those patients are attending to Kasr-Al Ainy Obstetrics outpatient clinic or casualty department during their 3rd trimester.

Ultrasound and doppler will be done to all patients to diagnose placenta accreta . The diagnosis will be confirmed by intraoperative assessments and histopathological examination of the uterus after cesarean hysterectomy

ELIGIBILITY:
Criteria:Inclusion Criteria

* Gestational age more than 28 weeks
* Single living fetus.
* One or more cesarean section or hysterotomy.
* Placenta previa (all grades) with high possibility of morbidly adherent placenta accreta (all types).

Exclusion Criteria:

* Maternal chronic medical disorder (diabetes mellitus or hypertension).
* Pregnancy induced disorders (pre-eclampsia or gestational diabetes).
* Associated fetal anomalies.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-05-22 (Estimated); Primary Completion 2018-08-22 (Estimated); Study Completion 2018-08-22 (Estimated)

PRIMARY OUTCOMES:
accuracy of ultrasound and doppler in detecting placenta accreta | 3 moths
  accuracy of uterine artery doppler in diagnosing placenta accreta diagnosed intraoperative or by histopathological examination done after cesarian hysterectomy

SECONDARY OUTCOMES:
accuracy of ultrasound in detecting placenta accreta diagnosed intraoperative or by histopathological examination done after cesarian hysterectomy | 3 months
  1. Loss of normal hypoechoic retroplacental zone
  2. Multiple vascular lacunae (irregular vascular spaces) within placenta
  3. Blood vessels or placental tissue bridging uterine-placental margin, myometrial-bladder interface, or crossing uterine serosa1
  4. Retroplacental myometrial thickness of 1 mm
  5. Bladder wall interruption
  6. Presence of placental bulge
  7. Utero-vesical hypervascularity
  3.Intraoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Hala Nabil, M.D, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided